CLINICAL TRIAL: NCT05880732
Title: The Effect of Preemptive Magnesium Sulfate on Postoperative Pain in Patients Undergoing Mastectomy
Brief Title: Magnesium Sulfate on Postoperative Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Ilknur Hatice Akbudak, MD, assistant professor doctor, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PAU123
Record Dates: First submitted 2023-04-05; First posted 2023-05-30 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Magnesium Sulfate

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Experimental): The study group (Group I) was given 50 mg/kg MgSO4 in 250 ml of isotonic 30 minutes before induction,
  Interventions: Drug: Magnesium Sulfate
- Group II (Placebo Comparator): the control group (Group II) was given only 250 ml of normal saline isotonic solution 30 minutes before induction,
  Interventions: Drug: normal saline isotonic solution

INTERVENTIONS:
Drug: Magnesium Sulfate — Magnesium sulfate (MgSO4) is an N-Methyl D-Aspartate (NMDA) receptor antagonist that has been used for postoperative analgesia and reducing both the duration and intensity of pain by preventing central sensitization in response to peripheral painful stimulus4-9.
  Arms: Group I
Drug: normal saline isotonic solution — only 250 ml of normal saline isotonic solution 30 minutes before induction,
  Arms: Group II

SUMMARY:
Breast cancer is the most diagnosed type of cancer in women in Turkey and in the world. According to the World Health Organization data, the rate of newly diagnosed breast cancer was reported as 11.6% in 20181. Acute postoperative pain occurs in 40% of patients undergoing surgery for breast cancer2. In the early postoperative period, opioids are commonly used analgesics in the treatment of pain, but they have various side effects such as gastrointestinal, urinary and respiratory symptoms3. Non-opioid analgesics can be used to reduce opioid use and thus limit its side effects. Magnesium sulfate (MgSO4) is an N-Methyl D-Aspartate (NMDA) receptor antagonist that has been used for postoperative analgesia and reducing both the duration and intensity of pain by preventing central sensitization in response to peripheral painful stimulus4-9. The primary aim of this study is to investigate the postoperative analgesic efficacy of MgSO4 in patients who were scheduled for mastectomy with the diagnosis of breast cancer. The secondary aim of our study is to evaluate the changes in perioperative vital signs that may occur due to MgSO4.

ELIGIBILITY:
Inclusion Criteria:

1. Female breast cancer patients scheduled for mastectomy and modified radical mastectomy
2. 18≥ years and
3. Patients with ASA score I-II

Exclusion Criteria:

1. The patient who refused the study
2. Drug allergy
3. Unregulated diabetes mellitus and hypertension
4. Cardiac failure with <45% ejection fraction
5. Renal failure (serum creatinine > 2 mg/dL)
6. Liver failure (blood transaminase values 2 fold higher than normal)
7. Glaucoma
8. Psychiatric or neurological disorders
9. Communication difficulties with patient
10. Calcium channel blockers or narcotic drugs uses before surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Postoperative pain was measured and recorded with the Verbal Numeric Rating Scale | 24 hours
  Postoperative pain was measured and recorded with the Verbal Numeric Rating Scale (VNRS) (0 no pain-10 very pain).

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale Univercity Medical School, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No